CLINICAL TRIAL: NCT04330664
Title: A Phase 1/2 Trial of MRTX849 in Combination With TNO155 in Patients With Advanced Solid Tumors With KRAS G12C Mutation KRYSTAL 2
Brief Title: Adagrasib in Combination With TNO155 in Patients With Cancer (KRYSTAL 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0017; CA239-0017 (Other: Bristol-Myers Squibb Protocol ID); 849-002 (Other: Mirati Therapeutics Protocol ID)
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancer; Metastatic Cancer; Malignant Neoplastic Disease
Keywords: KRAS G12C; Non-small cell lung cancer; Colorectal Cancer; Colon Cancer; Metastatic Cancer; Pancreatic Cancer; NSCLC; SHP2; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Dose Exploration (Experimental): Dose escalation of TNO155 to determine maximum tolerated dose of TNO155 in combination with MRTX849
  Interventions: Drug: MRTX849; Drug: TNO155
- Phase 1b Expansion (Experimental): Expansion cohort to ensure sufficient safety experience, pharmacokinetic information, and early evidence of clinical activity of MRTX849 in combination with TNO155 to recommend Phase 2 regimens
  Interventions: Drug: MRTX849; Drug: TNO155
- Phase 2 (Experimental): Separate cohorts of patients stratified by histological diagnosis for evaluation of clinical activity to evaluate clinical activity of MRTX849 and TNO155 in combination
  Interventions: Drug: MRTX849; Drug: TNO155

INTERVENTIONS:
Drug: MRTX849 — KRAS G12C Inhibitor
  Other Names: adagrasib
Drug: TNO155 — SHP2 Inhibitor

SUMMARY:
This study will evaluate the safety, tolerability, drug levels, molecular effects, and clinical activity of MRTX849 in combination with TNO155 in patients with advanced solid tumors that have a KRAS G12C mutation.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, pharmacokinetics, metabolites, pharmacodynamics, and clinical activity of MRTX849 in combination with TNO155 in patients with advanced solid tumors with a KRAS G12C mutation. MRTX849 is an orally available small molecule inhibitor of KRAS G12C and TNO155 is a selective, orally bioavailable allosteric inhibitor of wild-type SHP2.

This study was terminated prior to phase 2 initiating. Only phase 1 of the study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy with KRAS G12C mutation (phase 2 must be either Non-Small Cell Lung Cancer or Colorectal Cancer)
* Unresectable or metastatic disease
* No available treatment with curative intent
* Adequate organ function

Exclusion Criteria:

* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions likely to alter absorption of study treatment or result in inability to swallow
* Other active cancer
* Cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Characterize the safety of MRTX849 and TNO155 in patients having advanced solid tumor malignancies with KRAS G12C mutation. | 20 months
  Number of participants with treatment related adverse events
Evaluate the pharmacokinetics of MRTX849 and TNO155 | 20 months
  Blood plasma concentration

SECONDARY OUTCOMES:
Establish maximum tolerated dose | 12 months
  Number of participants with dose limiting toxicity
Evaluate clinical activity of MRTX849 | 20 months
  Objective response rate in accordance with Response Evaluation Criteria in Solid Tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (17):
  - Local Institution - 002-805, Los Angeles, California
  - Local Institution - 002-803, Orange, California
  - Local Institution - 002-828, Chicago, Illinois
  - Local Institution - 002-942, Wichita, Kansas
  - Local Institution - 002-804, Boston, Massachusetts
  - Local Institution - 002-808, Boston, Massachusetts
  - Local Institution - 002-811, Novi, Michigan
  - Local Institution - 002-809 D, City of Saint Peters, Missouri
  - Local Institution - 002-809 B, Creve Coeur, Missouri
  - Local Institution - 002-809 A, St Louis, Missouri
  - Local Institution - 002-809 C, St Louis, Missouri
  - Local Institution - 002-809, St Louis, Missouri
  - Local Institution - 002-809 E, St Louis, Missouri
  - Local Institution - 002-813, New York, New York
  - Local Institution - 002-806, New York, New York
  - Local Institution - 002-801, San Antonio, Texas
  - Local Institution - 002-810, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com